CLINICAL TRIAL: NCT02905955
Title: Negative Pressure Wound Management (NPWT) System for Inguinal Wounds After Venous Hybrid Procedures
Brief Title: Vacuumtherapy After Venous Hybrid Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL56603.068.16
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevena (Other)
  Interventions: Device: Prevena, KCI, Acelity, NPWT

INTERVENTIONS:
Device: Prevena, KCI, Acelity, NPWT — All patients will receive a Prevena NPWT (if inclusion criteria are met)

SUMMARY:
All patients with deep venous obstruction below the sapheno-femoral junction elective for hybrid procedure with creation of an arterio venous-fistula (AVF) in the MUMC or patients with primary percutaneous procedure (and thus venous obstruction above the sapheno-femoral junction) who present with occluded stents which need an additional AVF after thrombolysis will receive a Prevena NPWT. Incidence of wound infections and wound scoring will be performed afterwards.

ELIGIBILITY:
Inclusion Criteria:

* All patients with deep venous obstruction below the sapheno-femoral junction primary elective for hybrid procedure with creation of an AV-fistula in the MUMC
* Be able to communicate in Dutch
* Life expectancy >1 year

Exclusion Criteria:

* Patients with allergies for the components of the used negative pressure incision management system (Prevena)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With wound infections or Adverse Events That Are Related to Prevena incision management negative pressure wound therapy | 3 months
  Patients will be prospectively followed and checked for development of wound infections (grade 1-5). Therapy to treat the infections will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: J. Laanen, MD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided